CLINICAL TRIAL: NCT06873503
Title: Evaluation of the Effectiveness of the Weingart Plier in Combination With the Biting on Cotton Rolls in the Management of Pain During the Removal of Metal Brackets: A Randomized Controlled Trial
Brief Title: Assessment of Pain When Removing Metallic Brackets for Orthodontic Patients Using Two Removal Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-3-2025
Record Dates: First submitted 2025-03-07; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Orthodontic Appliance Complication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bracket removal with the mouth open (Active Comparator): Using a Weingart orthodontic plier, the patient will be asked to keep his mouth open during bracket removal.
  Interventions: Procedure: Bracket removal using a Weingart plier with the mouth open
- Bracket removal while biting on a cotton roll (Experimental): During bracket removal with a Weingart orthodontic plier, the patient will be asked to bite on a cotton roll between the upper and lower teeth.
  Interventions: Procedure: Biting on a cotton roll during brakcet removal

INTERVENTIONS:
Procedure: Bracket removal using a Weingart plier with the mouth open — The brackets will be removed using a Weingart plier. The patient will be asked to keep his mouth open during this procedure.
  Arms: Bracket removal with the mouth open
Procedure: Biting on a cotton roll during brakcet removal — The brackets will be removed using a Weingart plier. During this procedure, the patient will be asked to bite on a cotton roll.
  Arms: Bracket removal while biting on a cotton roll

SUMMARY:
Patients at the Orthodontic Department of the University of Damascus Dental School will be examined, and subjects who meet the inclusion criteria will be included. Then after finishing the orthodontic treatment, Patients were randomly assigned into two groups:

Open mouth group:

The debonding procedure was conducted using the open-mouth technique. All brackets were removed using a Weingart plier (American Orthodontics, Sheboygan, Wisc) by squeezing them from both sides of the mesial-distal surfaces. Before debonding, the stainless steel finishing archwires (0.017 × 0.025 inches) were removed.

Biting-on a-cotton-roll-group:

All brackets were removed using the same plier. The brackets were debonded using a Weingart plier (American Orthodontics, Sheboygan, Wisc) by squeezing them from both sides of the mesial-distal surfaces. Additionally, cotton rolls were placed between the upper and lower teeth, and patients were instructed to bite on them during the procedure. Before debonding, the stainless steel finishing archwires (0.017 × 0.025 inches) were removed. Patients in the second group were instructed to bite on a cotton roll throughout the debonding process.

DETAILED DESCRIPTION:
Pain is a subjective experience that can vary widely among individuals. It is influenced by several factors, including age, gender, personal pain threshold, psychological and social conditions, past negative experiences, and the degree of force applied.

Although various methods for bracket debonding, such as ultrasonic instrumentation, lasers, and electro-thermal debonding, are documented in the literature, hand tools like Weingart pliers remain among the most practical solutions. This study focused on using Weingart pliers to compare the pain scores in two techniques-open mouth and biting on a cotton roll-during bracket removal. These methods are widely used in orthodontic clinics and are readily available to orthodontists.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 16 to 25 years,
* Undergoing orthodontic treatment with MBT prescription 0.022-inch metal brackets with a single-mesh base (Pinnacle®, MBT compatible 0.022, OrthoTechnology™, Florida, USA) who were in the final stage of their treatment and planned for debonding,
* The brackets bonded with the same bonding cement (Ivoclar Heliosit Orthodontic Adhesive Composite) and the same primer (Ivoclar Vivadent Tetric N-Bond),
* Absence of debonded brackets at the debonding process,
* The 0.017 × 0.025-inch stainless steel finishing archwires in their places for at least one month,
* Good occlusal relationships and strong intercuspation,
* No recent use of medications such as painkillers or corticosteroids in the last day,
* Absence of acute or chronic dental pain induced by periodontal/periapical lesions or caries,
* There is an absence of a history of surgical treatment, including impacted tooth eruption, tooth transplantation, or the presence of mini-screws.

Exclusion Criteria:

* Presence of any craniofacial syndromes or systemic diseases
* Previous facial trauma
* Previous orthodontic treatment

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2024-05-19 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2025-01-05 (Actual)

PRIMARY OUTCOMES:
Perceived Pain Intensity | This assessment will be done once at the time of removing brackets (i.e., the patient will record the level of perceived pain within few seconds after removing each bracket for each tooth)
  Pain intensity will be evaluated using a 100-mm Visual Analog Scale (VAS), where a score of 0 indicates "no pain" and 100 indicated "extreme pain".
  Patients will be asked to record the perceived pain immediately after removing each bracket.
  This evaluation will cover all teeth on the upper and lower jaws.

CONTACTS AND LOCATIONS:
Overall Officials: Belal A. Drmch, DDS, Principal Investigator — Department of Orthodontics, Faculty of Dentistry, Damascus University, Damascus, Syria; Kinda Sultan, DDS MSc PhD, Study Director — Department of Orthodontics, Faculty of Dentistry, Damascus University
Locations (1):
- Department of Orthodontics, Faculty of Dentistry, University of Damascus, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karobari MI, Assiry AA, Mirza MB, Sayed FR, Shaik S, Marya A, Venugopal A, Alam MK, Horn R. Comparative Evaluation of Different Numerical Pain Scales Used for Pain Estimation during Debonding of Orthodontic Brackets. Int J Dent. 2021 Mar 4;2021:6625126. doi: 10.1155/2021/6625126. eCollection 2021. PMID 33747083
- [Background] Almuzian M, Rizk MZ, Ulhaq A, Alharbi F, Alomari S, Mohammed H. Effectiveness of different debonding techniques and adjunctive methods on pain and discomfort perception during debonding fixed orthodontic appliances: a systematic review. Eur J Orthod. 2019 Sep 21;41(5):486-494. doi: 10.1093/ejo/cjz013. PMID 30934051
- [Background] Gupta SP, Rauniyar S, Prasad P, Pradhan PMS. A randomized controlled trial to evaluate the effectiveness of different methods on pain management during orthodontic debonding. Prog Orthod. 2022 Mar 1;23(1):7. doi: 10.1186/s40510-022-00401-y. PMID 35229220
- [Background] Mangnall LA, Dietrich T, Scholey JM. A randomized controlled trial to assess the pain associated with the debond of orthodontic fixed appliances. J Orthod. 2013 Sep;40(3):188-96. doi: 10.1179/1465313313Y.0000000045. PMID 24009318
- [Background] Williams OL, Bishara SE. Patient discomfort levels at the time of debonding: a pilot study. Am J Orthod Dentofacial Orthop. 1992 Apr;101(4):313-7. doi: 10.1016/S0889-5406(05)80324-5. PMID 1558060